CLINICAL TRIAL: NCT02837354
Title: The Silent Cortical Infarcts in the Cerebral Amyloid Angiopathy: Is There a Link With Subarachnoid Hemorrhage?
Acronym: CAA
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: CAA
Record Dates: First submitted 2016-07-13; First posted 2016-07-19 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: CADASIL
Keywords: Cerebral Autosomal Dominant Arteriopathy with Subcortical Infarcts and Leukoencephalopathy
MeSH Terms: conditions — CADASIL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention

SUMMARY:
The Cerebral Amyloid angiopathy (CAA) is the leading cause of cortical hemorrhage after 65 years. The presence of cerebral infarction is also reported anatomically in the AAC. MRI studies of these infarcts are rare. They are described as punctate, cortical silent. Frequency and pathophysiology is poorly understood. The investigators put the question of a link with hemorrhagic lesions of the AAC.

DETAILED DESCRIPTION:
Main objective / secondary

The objectives are:

* To assess frequency of cortical infarcts in the cohort of patients recruited consecutively likely AAFC GHPSJ since 2007
* To assess the link between the presence of myocardial infarction and the clinical characteristics of patients and
* To study the relationship between topography and the brain hemorrhage one hand, meningeal hemorrhage other.

Inclusion / exclusion Any patient who was diagnosed as carrying a probable AAC according to the Boston criteria and has had a brain MRI with the following sequences: classic or enhanced diffusion (or DTI B2000), T1, T2 FLAIR, T2EG (T2 * or SWAN)

Methodology This is a non-interventional study single center, including AAC patients hospitalized in the Hospital Group Paris Saint-Joseph from May 2007 to May 2014.

Clinical patient characteristics were collected from their medical records. Patients are aware of the potential use of their data for medical research by information contained in the handbook of the institution.

Brain MRI will be proofread by a neurologist and a neuroradiologist to clarify:

* the number and location of myocardial puncture
* the number and location of macro-bleeding
* the number of microbleeds (micro-bleeding)
* the presence and location of subarachnoid hemorrhage and / or hemosiderosis
* the location of the puncture infarction compared to macro-hemorrhage and subarachnoid hemorrhage / hemosiderosis: ipsilateral <5cm, ipsilateral> 5cm, another location The clinical data and MRI will be entered on a file, with data anonymisation. Statistical analysis will be done by a neurologist service.

Number of topics:

* It is estimated that enrollment of patients with AAC by the UNV GHPSJ is approximately 10 patients per year. The number of screened patients during the study period should be about 70.
* Taking into account those whose MRI will be judged of insufficient quality (excluded), the number of patients included in the analysis should be around 50.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who was diagnosed as carrying a probable AAC according to the Boston criteria and has had a brain MRI with the following sequences: classic or enhanced diffusion

Exclusion Criteria:

* No conditions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient who was diagnosed as carrying a probable AAC according to the Boston criteria and has had a brain MRI with the following sequences: classic or enhanced diffusion
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2015-11 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
the number and location of myocardial puncture | Day 1
the number and location of macro-bleeding | Day 1
the number of microbleeds (micro-bleeding) | Day 1
the presence and location of subarachnoid hemorrhage and / or hemosiderosis | Day 1
the location of the puncture infarction | Day 1
  the location of the puncture infarction compared to macro-hemorrhage and subarachnoid hemorrhage / hemosiderosis: ipsilateral <5cm, ipsilateral> 5cm, another location

CONTACTS AND LOCATIONS:
Overall Officials: JOIN-LAMBERT Claire, MD, Principal Investigator — Groupe Hospitalier Paris Saint-Joseph (FRANCE)
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided